CLINICAL TRIAL: NCT04793308
Title: Comparison of Radicular Dentin Remaining, Risk of Perforation and Canal Transportation Between Manual Versus Rotary Instrumentation in Root Canals of Extracted Second Primary Molars: In Vitro Study
Brief Title: Radicular Dentin Remaining, Risk of Perforation and Canal Transportation in Manual Versus Rotary Instrumentation in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Associate Professor Dr. Rania Abdallah Nasr, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111120
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Root Canal Infection
Keywords: Deciduous teeth; pulpectomy; root canal preparation; canal transportation,; Cone Beam Computerized Tomography.

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1); (ProTaper Next, Rotary system). (Experimental): Group I teeth were prepared with rotary instrumentation using ProTaper Next (Dentsply, Switzerland)
  Interventions: Other: Endodontic files
- Group (2); K- files, Manual instruments. (Experimental): Group II root canals were prepared by manual instrumentation using K type files Mani, Japan).
  Interventions: Other: Endodontic files

INTERVENTIONS:
Other: Endodontic files — Engine-driven nickel titanium Ni-Ti instruments

SUMMARY:
Background: Root canal preparation techniques using manual instruments have found to be time-consuming and may lead to iatrogenic errors such as ledging, zipping, canal transportation, and apical blockage. To overcome this, much attention has been directed toward root canal preparation using nickel-titanium (NiTi)-rotary instruments. The flexibility and the instrument design of NiTi-rotary files allow it to closely follow the original root canal path. Aim: This in vitro study aims to compare the amount of dentin removal in primary molars instrumented with hand versus rotary files and the root canal transportation and risk of perforation using cone beam computed tomography (CBCT). Materials and Method: ( 20 ) extracted discarded mandibular second primary molars were selected to contribute in the study, having minimal apical resorption with presence of at least two-third remaining root structure with absence of visual perforating resorption. The teeth included in the study were stored in water or saline till the experimental time. The extracted primary molars were divided into two groups of the study: Group I was prepared with rotary instrumentation using ProTaper Next (Dentsply, Switzerland) and Group II was prepared by manual instrumentation using K type files. All the root canals (n=40) were prepared up to size 35 using the step-back technique. The teeth were subjected to CBCT scans for the evaluation of thickness of radicular dentin remaining, risk of perforation and canal transportation before and after instrumentation in the two groups at three different locations (2, 4 and 7 mm from the apex) . Dentin removal was calculated by superimposing images using the InVivo 5.1 software. Data were statistically analyzed using independent samples t test.

DETAILED DESCRIPTION:
Aim of the study:

To compare the shape & diameter of root canals, risk of perforation and the canal transportation after using rotary versus manual instruments on root extracted second primary molars.

Methodology:

Extracted second primary molars will be collected from the dental clinics of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.

The teeth are extracted either due to periodontal problems or because they are not restorable (beyond restoration) by the conventional coronal restorations or full coverage restorations in the case of root caries.

The teeth will be selected according to our inclusions and exclusion criteria. The teeth will be collected, sterilized and stored according to the Occupational Safety and Health Administration guidelines and regulations, ultrasonic scaler will be used to clean and remove soft tissue debris and calculus attached to the teeth.

Teeth will be divided into two groups:

Group (1); ((ProTaper Next, Rotary system). Group (2); K- files, Manual instruments. For cleaning and shaping of the canal system and mechanical preparation of root canal treatment.

Then shape of the canal (Canal transportation), canal diameter and risk of canal perforation will be compared in both groups.

Before and after preparation of the root canal, the shape of the canal will be assessed by using cone-beam computed tomography (CBCT) and diameter of the canal will be measured by using cone-beam computed tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* Extracted Second primary molars. Extracted second primary molars with at least 2/3 of root remaining or with minimal apical resorption.

Extracted second primary molars without visual perforation resorption.

Exclusion Criteria:

* Exfoliated second primary molars. If pre assessment radiograph for extracted second primary molars reveals internal or external root resorption.

Extracted second primary molars with extreme root curvature.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Radicular dentin remaining | 3 months
  Assessment of dentin remaining by Cone Beam Computerized Tomography (CBCT)
Transportation of Root Canal | 3 months
  Assessment of Root Canal Transportation by Cone Beam Computerized Tomography

SECONDARY OUTCOMES:
Risk of Perforation | 3 months
  By Cone Beam Computerized Tomography (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Assoc. Prof., Principal Investigator — Cairo University; Hany Sadek, Assoc. Prof., Principal Investigator — Cairo University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No